CLINICAL TRIAL: NCT03047434
Title: Characterization of Postoperative Pain in Shoulder Arthroscopy and Knee Arthroscopy and Assessment of the Defense and Veterans Pain Rating Scale for Persistent Post-Surgical Pain
Brief Title: Characterization of PostOp Pain in Shoulder and Knee Arthroscopy
Acronym: PurpleRain
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 413667
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The purpose of this study is to describe the chronology of post operative pain in patients undergoing total knee arthroplasty and total hip arthroplasty. Further, within this population the predictive validity of the Defense and Veterans Pain Rating Scale will be assessed for persistent post surgical pain.

DETAILED DESCRIPTION:
This is a prospective descriptive correlational design looking to characterize postoperative pain variables across various procedures that historically have significant levels of persistent post-surgical pain. Further, bivariate correlations at different time points will be examined to see how DVPRS along with Pain Assessment Screening Tool and Outcomes Registry (PASTOR) correlates with other measures.

Methodology/Technical Approach A total goal of 250 participants will be queried regarding their postoperative pain experience following shoulder arthroscopy and knee arthroscopy. Descriptive multidimensional tools (the DVPRS and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR)) will be used preoperative either during their preoperative surgical visit or the day of surgery and extending to 6 months postoperatively. As these tools have been utilized in previous studies for the prediction of persistent post surgical pain, the DVPRS will additionally be evaluated for its predictive validity as it is a short, easy-to-administer, bedside tool.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing the following surgeries: Total Knee Arthroscopy, Total Hip Arthroscopy.
2. DEERS eligible

Exclusion Criteria:

1. Younger than 18
2. Refuses participation
3. Cannot understand English
4. Has cognitive deficiencies
5. Ambulatory surgical status where they go home same day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Male and female military health care beneficiaries age 18 years and older presenting any of the following surgeries: total knee arthroplasty and total hip arthroplasty.
  2. The recruitment and participation in this study will have minimal impact on surrounding health care activities. This study is measuring pain in a more specific manner than usual to describe the perioperative pain experience and evaluate the predictive capability of the DVPRS. Measurements in this study will not be used to make therapeutic decisions. Participants will be screened from the Surgical Scheduling System (S3) and joint arthroplasty surgeon's scheduling nurse prior to surgery and approached upon their preoperative visit with their surgeon.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
To characterize the chronology/natural history of the postoperative pain experience in patients undergoing shoulder arthroscopy, knee, ankle arthroscopy in a multidimensional fashion from the immediate postoperative phase until 6 months post-surgery | 3-months and 6-months post-surgery
  Describe biopsychosocial functioning, as indicated by PROMIS domain scales and the DVPRS, at each time point, as well as longitudinal, polynomial data patterns for the aggregated sample.
  Examine whether longitudinal patterns vary according to surgical factors (e.g. procedure type, type of regional intervention received).
  Identify factors associated with low functioning and persistent opioid use at 3-months and 6-months post-surgery.
To assess the predictive validity of the DVPRS and PASTOR for persistent post-surgical pain at 3 and 6 months in patients undergoing the above surgical procedures. | 3-months and 6-months post-surgery
  ) When accounting for baseline levels, does postoperative Day 7 DVPRS scores predict persistent post- surgical pain at 3 months, as defined as 1 SD worse functioning on PROMIS Pain Interference? b) When accounting for baseline levels, does postoperative Day 7 DVPRS scores predict persistent post-surgical pain at 3 months, as defined as 1 SD worse functioning on PROMIS Neuropathic? c) What are the optimal cut-offs for the DVPRS at Day 7 in predicting persistent post-surgical pain at 3 months, as defined as 1 SD worse functioning on PROMIS Pain Interference?

CONTACTS AND LOCATIONS:
Overall Officials: Harold Gelfand, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- WRNMMC, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giordano NA, Kent M, Buckenmaier CC 3rd, Mauntel TC, Dickens JF, Millington M, Highland KB. A Longitudinal Comparison of Patient-Reported Outcomes Measurement Information System to Legacy Scales in Knee and Shoulder Arthroscopy Patients. Arthroscopy. 2021 Jan;37(1):185-194.e2. doi: 10.1016/j.arthro.2020.07.026. Epub 2020 Jul 25. PMID 32721547